CLINICAL TRIAL: NCT05763927
Title: Prospective Single-arm Phase II Clinical Study of Fruquintinib Combined With Toripalimab and SRT in Neoadjuvant Therapy for Locally Advanced Rectal Cancer
Brief Title: Neoadjuvant Therapy for Locally Advanced Rectal Cancer With Fruquintinib, Toripalimab and SRT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yaqin Zhao, Associate Chief Physician, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-013-CH11 IIT-CR
Record Dates: First submitted 2023-02-27; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Rectal Cancer
Keywords: Fruquintinib; Toripalimab; SRT; neoadjuvant therapy; pCR
MeSH Terms: conditions — Rectal Neoplasms | interventions — HMPL-013; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fruquintinib& Toripalimab& SRT (Experimental): Induction treatment:
  Fruquintinib 5mg d1-d14； Toripalimab 240 mg intravenously d1；
  Consolidation treatment:
  SRT: 25 Gy in 5 fractions d22-d26； Fruquitinib 5mg d22-d35，43-56,64-77； Toripalimab 240 mg intravenously d22、43、64；
  Surgery: Surgical resection will be performed according to the principles of TME(total mesorectal excision) 2-4 weeks after the last dose administration of Fruquintinib；
  Adjuvant chemotherapy: Standard chemotherapy or observation according to the judgement of Principle Investigator and patients' willing.
  Interventions: Drug: Fruquintinib; Drug: Toripalimab; Radiation: Short-course radiotherapy; Procedure: TME

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib 5mg 2w on/1w off, 21d/cycle, totally 4 cycle.
Drug: Toripalimab — Toripalimab 200mg d1, 21d/cycle, totally 4 cycle.
Radiation: Short-course radiotherapy — 25 Gy in 5 fraction, d22-26.
  Other Names: SRT
Procedure: TME — Surgical resection of the primary tumour in the rectum, 2-4weeks after the last dose of fruquintinib
  Other Names: Total mesorectal excision

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of combined fruquintinib、toripalimab and SRT in neoadjuvant therapy for locally advanced rectal cancer.

DETAILED DESCRIPTION:
The aim of this study is to investigate whether combined fruquintinib、toripalimab and SRT can achieve breakthrough efficacy in neoadjuvant therapy for locally advanced rectal cancer, achieving a better pCR rate and better tolerance compared with conventional neoadjuvant therapy for locally advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Rectal adenocarcinoma was confirmed pathologically;
2. Baseline clinical staging was T3-4 and/or N+, and rectal enhanced MRI was recommended as staging standard;
3. distance from anus ≤12cm;
4. No distant metastasis;
5. Age 18-70, regardless of gender;
6. ECOG(Eastern Cooperative Oncology Group) score ≤1;
7. No chemotherapy or other anti-tumor therapy was used before inclusion;
8. Major organ functions within 28 days prior to treatment meet the following criteria: A. Blood routine examination criteria (within 14 days without blood transfusion) : Hemoglobin (HB) ≥80g/L, absolute value of neutrophil (ANC) ≥1.5×109/L, absolute value of lymphocytes ≥ the lower limit of normal value, platelet (PLT) ≥80×109/L; B. Biochemical tests should meet the following criteria: Total bilirubin (TBIL) ≤1.5 times the upper limit of normal value (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN; C. Coagulation tests should meet the following standards: International standardized ratio (INR) or prothrombin time (PT) ≤1.5 ULN; Activated partial thrombin time (APTT) ≤1.5 ULN (if the patient is on anticoagulant therapy, as long as PT and APTT are within the expected treatment range); D. Thyroid function: T3 and T4 levels were normal after drug treatment;
9. No history of autoimmune diseases or current autoimmune diseases;
10. Subjects must give informed consent to the study prior to the study and have voluntarily signed a written informed consent;
11. The subjects can communicate well with the researcher and complete the study according to the protocol; Women of reproductive age ;
12. should agree to use contraception (such as an intrauterine device, birth control pill or condom) during the study period and 120 days after the end of the study; Serum or urine pregnancy tests were negative during the 7 days prior to study enrollment.

Exclusion Criteria:

1. Patients who have previously received immune checkpoint inhibitors;
2. Known allergic reactions to PD-1 monoclonal antibody active ingredients, TKI inhibitor-related ingredients or any excipients;
3. Patients with organ bleeding or bleeding tendency, except for rectal primary tumor bleeding (need investigator to assess the risk of bleeding;
4. Pregnant or lactating women;
5. years or at the same time have a history of other malignant tumors, but cured skin basal cell carcinoma and cervical carcinoma in situ and thyroid;
6. Patients with uncontrolled epilepsy, central nervous system disease or mental disorders, the investigator judged that their clinical severity may hinder the signing of informed consent or affect the patient 's compliance with oral drugs;
7. Clinically serious (i.e., active) heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) class II or more severe congestive heart failure or severe arrhythmia requiring drug intervention, or a history of myocardial infarction within the last 12 months;
8. Subjects requiring systemic treatment with corticosteroids (greater than 10 mg prednisone equivalent daily) or other immunosuppressive agents (including organ transplant recipients) within 2 weeks before the first dose of study drug;
9. Participated in other interventional drug clinical trials within 4 weeks before the first dose;
10. Major surgery or severe trauma within 4 weeks before the first dose of study drug;
11. Serious infection (CTCAE greater than grade 2) within 4 weeks before the first dose of study drug,Such as severe pneumonia, bacteremia, infectious complications requiring hospitalization; baseline chest imaging suggests active pulmonary inflammation, symptoms and signs of infection within 2 weeks before the first dose of study drug, or the need for oral or intravenous antibiotics (excluding prophylactic antibiotics);
12. Active autoimmune diseases, history of autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases and syndromes); autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormone, using stable doses of insulin type 1 diabetes can be included; but excluding vitiligo or recovered childhood asthma/allergy, without any intervention in adults;
13. History of immunodeficiency, including positive HIV test, or other acquired, congenital immunodeficiency diseases, or history of organ transplantation and bone marrow transplantation;
14. Active pulmonary tuberculosis infection found by medical history or CT examination, Or patients with a history of active pulmonary tuberculosis infection within 1 year before enrollment, or patients with a history of active pulmonary tuberculosis infection but without regular treatment 1 year before enrollment;
15. Subjects with active hepatitis (HBV DNA ≥ 2000 IU/ml or 10000 copies/ml), hepatitis C (hepatitis C antibody positive,HCV-RNA was above the lower limit of detection of the assay);
16. Had a known history of psychotropic drug abuse, alcoholism, or drug use;
17. Had a history, illness, treatment, or laboratory abnormality that could interfere with the results of the trial, prevent the subject from participating throughout the study, or the investigator considered participation to be in the subject 's best interest.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
pCR following neoadjuvant chemotherapy | approximately 2 weeks after the resection of primary lesion
  Pathologic complete response (pCR) rate defined as number of participants out of total that had no residual invasive disease (malignant cells)

SECONDARY OUTCOMES:
R0 resection rate | approximately 2 weeks after the resection of primary lesion
  number of R0 surgery divide all participants (44pts)
Objective response rate | approximately before the resection of primary lesion
  Objective tumour response (ORR) will is defined as the proportion of subjects who achieve a partial or complete response according to RECIST criteria version 1.1
1 year DFS(disease free survival) rate | 1 year
  evaluate the 1-year DFS rate after the resection of primary lesion（only patients who acquire R0 resection）
1 year OS(overall survival) rate | 1 year
  evaluate the 1-year OS rate after the neoadjuvant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Shared for: scientific research institutions, academic journal Shared for: scientific research institutions, academic journal, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
IPD(individual patient data) Sharing Plan:
  Shared for: scientific research institutions, academic journal editors, government agencies Sharing conditions: IPD sharing shall meet the following conditions: Requestor must provide study agreement and relevant ethical review committee approval documents Requestor must ensure legality of data use and privacy protection Requestor must agree to data sharing, and the study team has the right to review the Requestor 's study plan and provide necessary support and interpretation of data
  Scope of shared data: The shared data includes ECG and clinical data of all subjects, but excluding personal information of subjects
Time Frame: Sharing period is 5 years, which start from one year after primary outcome publication.
Access Criteria: Shared for: scientific research institutions, academic journal editors, government agencies Sharing conditions: IPD sharing shall meet the following conditions: Requestor must provide study agreement and relevant ethical review committee approval documents Requestor must ensure legality of data use and privacy protection Requestor must agree to data sharing, and the study team has the right to review the Requestor 's study plan and provide necessary support and interpretation of data